CLINICAL TRIAL: NCT06778551
Title: Effectiveness of an Exercise Program Focused on the Thoracic Spine, Scapular Region, and Shoulder in Patients With Subacromial Impingement: A Multicenter Prospective Randomized Controlled Study
Brief Title: Shoulder School: A Multicenter Prospective Randomized Controlled Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sandra Jiménez-del-Barrio (Other)
Collaborators: Sanidad de Castilla y León (Other)
Responsible Party: Sponsor-Investigator, Sandra Jiménez-del-Barrio, PhD. Sandra Jiménez del Barrio, University of Valladolid
Organization: University of Valladolid (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REF CEIm 3200
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-01

CONDITIONS: Subacromial Impingement Syndrome
Keywords: quality of life; Subacromial impingement syndrome; pain; exercise
MeSH Terms: conditions — Shoulder Impingement Syndrome; Pain; Motor Activity | interventions — Exercise; Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (Experimental): A therapeutic exercise protocol will be carried out, consisting of 2 sessions per week for 8 weeks, supervised and guided by a physiotherapist. The objective is to improve thoracic mobility, as well as the strength and motor control of the scapular retractor and protractor muscles (middle and lower trapezius, rhomboids, and serratus anterior) and the rotator cuff.
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION
- Control group (Active Comparator): The protocol will include the application of therapeutic ultrasound. For this application, ultrasound gel will be used to reduce friction and improve the transmission of waves. Using a 5 cm² transducer, pulsed ultrasound will be applied at a frequency of 3 MHz and an intensity of 1 W/cm² for 10 minutes. Patients will be informed that they should not feel any sensation during the procedure, and if they do, the intensity will be reduced. Finally, kinesitherapy will be applied through classic shoulder mobility exercises.
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — A therapeutic exercise protocol will be carried out, consisting of 2 sessions per week for 8 weeks, supervised and guided by a physiotherapist. The objective is to improve thoracic mobility, as well as the strength and motor control of the scapular retractor and protractor muscles (middle and lower trapezius, rhomboids, and serratus anterior) and the rotator cuff.
  Arms: Exercise group
Other: Control (Standard treatment) — The protocol will include the application of therapeutic ultrasound. For this application, ultrasound gel will be used to reduce friction and improve the transmission of waves. Using a 5 cm² transducer, pulsed ultrasound will be applied at a frequency of 3 MHz and an intensity of 1 W/cm² for 10 minutes. Patients will be informed that they should not feel any sensation during the procedure, and if they do, the intensity will be reduced. Finally, kinesitherapy will be applied through classic shoulder mobility exercises.
  Arms: Control group

SUMMARY:
Subacromial impingement syndrome (SIS) is the most common cause of shoulder pain. Patients with SIS present with localized shoulder pain, sometimes nocturnal, which leads to a decrease in shoulder strength and function, significantly affecting their quality of life. Several authors have proposed that reduced scapular movement could be a direct causal mechanism for the symptoms associated with SIS. There is evidence supporting the benefits of passive techniques applied to the scapula and thoracic spine in terms of symptom relief and improved function.

The high healthcare demand from patients with SIS, combined with long waiting lists in physiotherapy, rehabilitation, and trauma services related to this dysfunction, underscores the need for a group-based therapeutic exercise strategy.

Objective To analyze the effects of a shoulder school program led by a physiotherapist and based on therapeutic exercise focused on active scapular and thoracic work, compared to conventional treatment in patients with SIS referred to Primary Care Physiotherapy Units (UFAP), regarding pain, functional capacity, and quality of life.

Methods Design: Single-blind, multicenter, prospective, randomized, controlled non-inferiority study.

Sample: Patients with SIS referred to UFAP. Dependent Variables: Pain, functional capacity, quality of life, joint mobility, scapular function, and patient satisfaction.

Independent Variables:

Intervention group: Shoulder school program including exercises focused on scapular, thoracic, and rotator cuff function.

Control group: Conventional physiotherapy treatment. Randomization: Cluster randomization by centers. Analysis: Data will be analyzed using SPSS version 25.0.

Clinical Implications This study will provide objective data on the effects of implementing a group exercise program guided by a physiotherapist. The results could offer evidence for a resource that may be highly useful in Primary Care Physiotherapy. This approach has the potential to optimize labor, time, and space resources within this healthcare service.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old
* Shoulder pain lasting more than 6 weeks, attributable to rotator cuff tendinopathy or tendinosis, subacromial impingement syndrome, or subacromial pinching, according to the diagnostic criteria of the British Shoulder and Elbow Society. Must meet 2 of the following criteria: painful arc during flexion or abduction, positive Neer test, positive Hawkins-Kennedy test, or pain with resisted movement of external rotation, abduction, or positive Jobe test.
* Ability to understand and complete the evaluation questionnaires

Exclusion Criteria:

* History of significant shoulder trauma (fractures, dislocations, complete tears requiring surgery)
* Neurological disorders affecting the shoulder
* Other severe shoulder pathologies (inflammatory arthritis, frozen shoulder, or glenohumeral instability)
* Received corticosteroid injections or physical therapy for the shoulder in the last 6 months
* Referred to another specialized care service, such as surgery, due to SIS
* Pregnancy
* BMI (Body Mass Index) greater than 30 kg/m².

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Pain intensiy | From enrollment to the end of treatment at 8 weeks
  Visual analogue scale is a subjective pain intensity measurement tool in which subjects are asked to indicate their perceived pain intensity on a 10 cm line. Patients will be informed that the left end of the scale represents "no pain" and the right end represents "the worst pain imaginable." It will be explained that marking closer to the right corresponds to a higher score (10 cm) and greater pain, while marking closer to the left corresponds to a lower score (0 cm) and a better state of health.
Physical Function | From enrollment to the end of treatment at 8 weeks
  The SPADI (Shoulder Pain and Disability Index) is a questionnaire used to measure shoulder symptoms and function. It consists of 13 questions divided into two categories: pain and activity limitation. It is a self-administered questionnaire where patients respond to the questions using a visual analog scale. A higher score on the questionnaire indicates greater pain and greater restriction in activities.

SECONDARY OUTCOMES:
Disability | From enrollment to the end of treatment at 8 weeks
  The DASH is one of the most commonly used questionnaires to assess symptoms and function of the upper extremity. This questionnaire considers the level of difficulty experienced in performing physical activities due to upper limb problems and the severity of symptoms. It consists of 30 items divided into three sections: 11 general questions, 4 related to work, and 4 related to sports. Each item offers 5 response options, ranging from 1 (representing no difficulty) to 5 (representing complete inability to perform the activity).
Quality of life | From enrollment to the end of treatment at 8 weeks
  WORC Questionnaire (Western Ontario Rotator Cuff Index) is a questionnaire designed to assess the impact of treatment on quality of life in relation to rotator cuff dysfunction. It includes 21 items covering physical symptoms, sports and recreational activities, work-related activities, lifestyle, and emotional aspects.
Scapular stability | From enrollment to the end of treatment at 8 weeks
  The lateral scapular slide test is a functional assessment that measures scapular mobility in different arm positions. This test evaluates the distance between the inferior angle of the scapula and the corresponding spinal spinous process. It is performed in three positions: arms at the sides of the body, hands on the waist, and shoulders at 90° in internal rotation.
Global rating score | At the end of treatment at 8 weeks
  Global Rating of Change (GROC Scale) is a 15-item scale that assesses the clinical significance that the patient assigns to their outcomes. It allows for the evaluation of the therapeutic value of the proposed techniques.
Shoulder Joint Mobility | From enrollment to the end of treatment at 8 weeks
  The painless active range of motion will be measured using a digital inclinometer during flexion, abduction, and internal and external rotation movements.
Isometric muscle strength | From enrollment to the end of treatment at 8 weeks
  The strength of internal and external rotation will be assessed with the shoulder at 90º of abduction.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Soria, Soria, Spain

IPD SHARING:
Plan to Share IPD: No